CLINICAL TRIAL: NCT07031791
Title: PETRA: Pictorial Assessment of Task Occurrence and Upper Limb Avoidance Behaviors
Acronym: PETRA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0163
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Thoraco-brachial Outlet Syndrome; ADAP-shoulder Scale; PETRA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with thoraco-brachial outlet syndrome: PETRA questionnaire
  Interventions: Other: PETRA questionnaire

INTERVENTIONS:
Other: PETRA questionnaire — The questionnaire is given to the patient to complete in the waiting room. The completed questionnaire is given to the doctor at the end of the consultation.

SUMMARY:
The clinical evaluation of patients suspected of having thoracic brachial outlet syndrome (TBS) is not standardized, as it may be for the lower limbs. Assessment of symptoms and functional impact is based on questionnaires (Disability of the Arm, Shoulder and Hand: DASH, Short Form 36: SF36, Mobility of the Arm and Shoulder: MASC, Thoracic and Upper limb ischemia Pain: TULIP), which are complex to complete, sometimes non-lateralized, and do not take into account the frequency of occurrence of certain gestures or the avoidance behaviours adopted by patients.

For avoidance behaviors, a recent tool has been proposed in the form of the Avoidance Daily Activities Photo Scale (ADAP shoulder scale). However, this questionnaire has not been translated into French and does not reflect the frequency with which patients are confronted with the different tasks proposed.

The aim of this study is to test the feasibility of a new questionnaire (PETRA), derived from the ADAP-shoulder scale, which is simple for patients to complete, quick to analyze and calculable directly by the doctor, and suitable for the general population, whether for initial assessment or follow-up.

The PETRA aims to assess avoidance behaviours in the face of daily tasks, but also the frequency of occurrence of these tasks in order to evaluate a disabling score that weights the avoidance index according to the degree of exposure to the proposed tasks.

The investigators hypothesize that the PETRA questionnaire could eventually be used routinely.

ELIGIBILITY:
Inclusion Criteria:

* Adult,
* Person referred for suspected TDSB

Exclusion Criteria:

* Person unwilling to complete questionnaire and participate,
* Person unable to understand the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for thoraco-brachial outlet syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
PETRA questionnaire | Inclusion
  The questionnaire enables patients to indicate the extent to which they avoid performing everyday tasks, based on 15 questions taken from the ADAP Shoulder Scale, to which have been added five questions on the ability to pull an object, throw an object and dry oneself. Each question is on a numerical scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No